CLINICAL TRIAL: NCT02811497
Title: An Open-label, Phase II Basket Study of a hypoMEThylating Agent Oral Azacitidine and DURvalumab (MEDI4736) (Anti-PDL1) in Advanced Solid Tumors (METADUR)
Brief Title: Study of Azacitidine and Durvalumab in Advanced Solid Tumors
Acronym: METADUR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: METADUR-001
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Microsatellite Stable Colorectal Carcinoma; Platinum Resistant Epithelial Ovarian Cancer Type II; Estrogen Receptor Positive and HER2 Negative Breast Cancer
MeSH Terms: interventions — Azacitidine; cc-486; durvalumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azacitidine and Durvalumab (Experimental): Azacitidine will be given by mouth at a fixed dose of 300 mg daily for 14 consecutive days of every 28 day cycle for 3 cycles.
  Durvalumab will be given intravenously (by vein) at a fixed dose of 1500 mg (over 1 hour) on Day 1 of every 28 day cycle for 12 months or until disease progression.
  Interventions: Drug: Azacitidine; Drug: Durvalumab

INTERVENTIONS:
Drug: Azacitidine
  Other Names: CC-486
Drug: Durvalumab

SUMMARY:
This is a phase 2 study of investigational drug, durvalumab given in combination with azacitidine (CC-486). The main purpose of this phase 2 study is to assess the antitumor activity of azacitidine in combination with durvalumab patients with microsatellite stable colorectal carcinoma (MSS-CRC), platinum resistant epithelial ovarian cancer type II (PR-OC), and estrogen receptor positive and HER2 negative breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent.
* Age ≥18 years or ≥20 years for Japanese participants.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
* Life expectancy of ≥12 weeks
* Have histologically or cytologically-documented, locally-advanced, or metastatic solid malignancy that is incurable and has either (a) failed prior standard therapy, (b) for which no standard therapy exists, or (c) standard therapy is not considered appropriate by the patient and treating physician.
* Have one of the following advanced (unresectable and/or metastatic) solid tumor indications:

  * Microsatellite Stable Colorectal Carcinoma (MSS-CRC)
  * Platinum Resistant Epithelial Ovarian Cancer Type II (PR-OC)
  * Estrogen Receptor Positive and HER2 Negative Breast Cancer (ER+/HER2- BC):
* The following considerations will be made regarding prior treatment regimens:

  * MSS-CRC: must have progressed or be intolerant of 5-FU, irinotecan, oxaliplatin and epidermal growth factor receptor (EGFR) mAb in patients with RAS wild type tumors, in recurrent/metastatic setting.
  * PR-OC: must have progressed on at least 1, maximum of 2 lines of cytotoxic agents in the platinum resistant disease setting
  * ER+/HER2- BC: must have progressed on at least 2, maximum of 5 lines of cytotoxic agents in recurrent/metastatic setting.
* Adequate normal organ and marrow function
* Willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up.
* At least one measurable lesion according to RECIST v1.1.
* At least one lesion safely accessible for biopsy.
* Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion.
* Consent to provide archival tumor tissue (initial and subsequent tumor biopsy samples, if possible) for correlative biomarker studies, if available.
* Female subject of childbearing potential1 should have two negative pregnancy tests as verified by the investigator prior to starting any investigational product therapy
* Females of childbearing potential who are sexually active with a non-sterilized male partner must agree to practice true abstinence or use at least two effective methods of contraception for the study defined period.
* Non-sterilized males who are sexually active with a female partner of childbearing potential must agree to use at least two effective methods of contraception for the study defined period.

Exclusion Criteria:

* Involvement in the planning and/or conduct of the study or previous enrolment in the present study.
* Participation in another clinical study with an investigational product during the last 28 days or 5 half-lives prior to study Day 1. Concurrent enrolment in an observational (noninterventional) clinical study or the follow-up period of an interventional study is allowed.
* Any previous treatment with a PD1 or PD-L1 inhibitor, including durvalumab. Prior anti-CTLA4 agents are allowed. Prior therapy with T-cell co-stimulatory agents (e.g. anti-CD137 antibody, anti-OX40 antibody) are allowed.
* Prior therapy with CC-486, azacitidine, decitabine or any other hypomethylating agent.
* History of another primary malignancy with exceptions.
* Receipt of the last dose of anti-cancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies, other investigational agent) ≤ 28 days prior to the first dose of study drug (and within 6 weeks for nitrosourea or mitomycin C).
* Mean QT interval corrected for heart rate (QTc) ≥470 ms.
* Current or prior use of immunosuppressive medication within 28 days before the first dose of durvalumab with exceptions.
* Any unresolved toxicity CTCAE grade 2 from previous anti-cancer therapy.
* Any prior Grade ≥3 immune-related adverse event (irAE) while receiving any previous immunotherapy agent, or any unresolved irAE >Grade 1, with exception of chronic endocrinopathy that is stable on hormone replacement.
* Active or prior documented autoimmune disease within the past 2 years.
* Active or prior documented inflammatory bowel disease (e.g., Crohn's disease, ulcerative colitis).
* History of primary immunodeficiency
* History of allogeneic organ transplant
* History of hypersensitivity to study drug formulations, including azacitidine, mannitol, or durvalumab, its constituents, or to any other humanized monoclonal antibody
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, active peptic ulcer disease or gastritis, active bleeding diatheses including any patient known to have evidence of acute or chronic hepatitis B, hepatitis C or human immunodeficiency virus (HIV), or psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent
* Known history of previous clinical diagnosis of tuberculosis
* Receipt of live attenuated vaccination within 30 days prior to study entry or within 30 days of investigational products.
* Female patients who are pregnant, breast-feeding or male or female patients of reproductive potential who are not employing an effective method of birth control.
* Irritable bowel syndrome or other serious gastrointestinal chronic conditions associated with diarrhea within the past 3 years prior to the start of treatment, and/or history of prior gastrectomy or upper bowel removal, or any other gastrointestinal disorder or defect that would interfere with the absorption, distribution, metabolism or excretion of the investigational product and/or predispose the patient to an increased risk of gastrointestinal toxicity.
* Untreated central nervous system (CNS) metastatic disease, leptomeningeal disease, or cord compression.
* Patients with uncontrolled seizures.
* Any concurrent chemotherapy, immunotherapy, or biologic or hormonal therapy for cancer treatment with the exception of patients on adjuvant endocrine therapy for a history of non-invasive breast cancer.
* Major surgery within 28 days prior to Day 1 of the study or still recovering from prior surgery.
* Any condition that, in the opinion of the investigator, would interfere with evaluation of study treatment or interpretation of patient safety or study results.
* Patients who are involuntarily incarcerated or are unable to willingly provide consent or are unable to comply with the protocol procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-09; Primary Completion 2018-11-08 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Overall response rate (ORR) | 4 weeks

SECONDARY OUTCOMES:
Disease Control Rate (DCR) | 16 weeks
Progression-free survival (PFS) | 5 years
Overall survival (OS) | 5 years
Incidence of treatment-emergent adverse events (AEs) | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Lillian Siu, M.D., Principal Investigator — Princess Margaret Cancer Centre
Locations (1):
- Princess Margaret Cancer Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Taylor K, Loo Yau H, Chakravarthy A, Wang B, Shen SY, Ettayebi I, Ishak CA, Bedard PL, Abdul Razak A, R Hansen A, Spreafico A, Cescon D, Butler MO, Oza AM, Lheureux S, Stjepanovic N, Van As B, Boross-Harmer S, Wang L, Pugh TJ, Ohashi PS, Siu LL, De Carvalho DD. An open-label, phase II multicohort study of an oral hypomethylating agent CC-486 and durvalumab in advanced solid tumors. J Immunother Cancer. 2020 Aug;8(2):e000883. doi: 10.1136/jitc-2020-000883. PMID 32753546